CLINICAL TRIAL: NCT01515982
Title: Physical Exercise as an Additional Treatment for Alzheimer Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Jerson Laks, Principal investigator, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60liv02-09B
Record Dates: First submitted 2012-01-12; First posted 2012-01-24 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; Aerobic exercise; Physical training; Cognitive function; Functional capacity.
MeSH Terms: conditions — Alzheimer Disease | interventions — Exercise; Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic exercise (Experimental): The training exercise intensity is established at 60% of VO2máx. Each aerobic session began with a 10-minute warm-up period (40%VO2máx), followed by 20 minutes of continuous treadmill walking at an intensity established by 60% of VO2máx. The exercise session will be concluded with a 5 minutes of cool down. Heart hate (Polar® Sport Tester, Finland) and perceived exertion (Borg Scale) will be monitored and recorded at each five minutes during each exercise session by physical education instructors.
  Interventions: Behavioral: Aerobic Exercise; Behavioral: Control Group
- Control group (No Intervention): All participants were asked not to commence any new exercise regimen.

INTERVENTIONS:
Behavioral: Aerobic Exercise — The training exercise intensity is established at 60% of VO2máx. This intensity was determined using exercise prescription guidelines established by the American College of Sports Medicine (ACSM). Each aerobic session began with a 10-minute warm-up period (40%VO2máx), followed by 20 minutes of continuous treadmill walking at an intensity established by 60% of VO2máx. The exercise session will be concluded with a 5 minutes of cool down. Heart hate (Polar® Sport Tester, Finland) and perceived exertion (Borg Scale) will be monitored and recorded at each five minutes during each exercise session by physical education instructors.
  Arms: Aerobic exercise
Behavioral: Control Group — All participants were asked not to commence any new exercise regimen.
  Arms: Aerobic exercise

SUMMARY:
The state of the art with regard to the neurodegenerative dementias, especially for Alzheimer´s disease (AD), is that their progression is still irreversible causing cognitive, motor, and behavioral impairment. Although the current pharmacological treatments attenuate cognitive decline in some cases, the majority of treatments does not avoid the motor and functional changes caused by the progress of the disease. Although several studies show that exercise has a positive effect when it comes to the treatment of the disease, some methodological questions affect the application of the training protocols. The use of recognized intensity patterns like maximum oxygen uptake (VO2max) and maximum heart rate (HRmax) percentage to control the training of patients with dementia is still rare in the literature. Therefore, this seems to interfere on the definition of an ideal prescription. Following this line of reasoning, the purpose of the present study is to assess the effect of moderate aerobic exercise on cognition and functional abilities in AD patients. Design: Randomized controlled trial, double-blinded, with 16-week follow-up. Setting: Center for Alzheimer's disease in the Institute of Psychiatry of the Federal University of Rio de Janeiro. Participants: Elderly with Alzheimer disease. Interventions: The patients will be randomly assigned to an exercise group (EG) on a treadmill (30 minutes, twice a week and moderate intensity of 60% VO2max) and a control group (CG). Main outcome measures: Cognitive function will be assessed using CAMCOG, Trail Making Test A, Digit Span, Stroop Test, Rey auditory-verbal learning test and Clock Test, and functional capacity will be evaluated using Berg Balance Scale (BERG), Sit-to-Stand test (STS), functional reach test (FR), and the time to up and go test (TUGT).

DETAILED DESCRIPTION:
* Design: Four-month controlled, randomized, and double-blind study. The patients will be recruited by trained psychiatrists from the Center for Alzheimer's disease in the Institute of Psychiatry of the Federal University of Rio de Janeiro (IPUB/UFRJ). They will be randomized with a blind design to an exercise group (EG) and control group (CG) by a researcher who will not participate of the initial assessments.
* Intervention

On completion of the baseline assessment, all patients will be invited to engage in the exercise program. Those who accept to take part and will be available, having easy access to the facilities, will be included in the sample. The other ones will be included in the control group. So, subjects will be divided by two groups: medical care (control) and medical care + physical exercise.

1. Medical care control group (C): Subjects will maintain clinical treatment.
2. Medical care + exercise group (E): This group will be prescribed the exercise treatment as an adjunctive intervention to drug therapy. Patients who accept to participate in this group will be evaluated with a thorough clinical exam and with a resting electrocardiogram. The training exercise intensity is established at 60% of VO2máx. This intensity was determined using exercise prescription guidelines established by the American College of Sports Medicine (ACSM). Each aerobic session began with a 10-minute warm-up period (40%VO2máx), followed by 20 minutes of continuous treadmill walking at an intensity established by 60% of VO2máx, according to ACMS guidelines (2006). The exercise session will be concluded with a five minutes of cool down. Heart hate (Polar® Sport Tester, Finland) and perceived exertion (Borg Scale) will be monitored and recorded at each five minutes during each exercise session by physical education instructors. Subjects will be encouraged to attend two supervised exercise sessions per week for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer Disease according to the National Institute of Neurological and Communicative Disorders and Stroke- Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) and National Institute of Neurological Disorders and Stroke- Association Internationale pour la Recherche et l' Enseignement en Neurosciences (NINDS-AIREN),respectively
* Mini-Mental State Examination (MMSE) score ≥ 15
* Clinical Dementia Rating (CDR) score 1
* Regular use of anticholinesterase drugs for at least six months
* Cardiologist's authorization
* At least six months without practicing physical exercises.

Exclusion Criteria:

* Clinical depression or Cornell Scale ≥ 7
* Other types of dementia
* Physical limitation due to other pathologies or associated neurological disease
* Severe or uncontrolled arterial hypertension
* Marked visual and/or auditory deficit
* Incapacity to perform physical exercise due to neurological or neuromuscular impairments
* Illiteracy
* Less than six months of treatment at the outpatient unit.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in CAMCOG scale at 16 weeks | from date to randomization at 16 weeks
  The general cognitive state will be assessed by the Brazilian validated version of the CAMCOG, which is part of the cognitive evaluation developed by the CAMDEX (Cambridge Examination for Mental Disorders of the Elderly) and is subdivided in scales which assess orientation, expressive and comprehensive language, memory (including remote memory, recent memory and learning processes), attention, praxis, calculation, abstract thinking and perception.

SECONDARY OUTCOMES:
Change from baseline in Time to Up and Go Test at 16 weeks | from date to randomization at 16 weeks
  The "Timed Up and Go" test (TUGT) and its modified version "Modified Timed up and go" (TUG mod) have been used with the objective of evaluating the functional mobility and the double task, respectively. In the first test, the patient walks three meters while the time is counted, and, in the second one, the patient is asked to walk and evoke names of animals. More than 10 seconds is considered risk of functional loss.
Change from baseline in Sit-to-Stand test at 16 weeks | from date to randomization at 16 weeks
  The Sit-to-Stand test (STS) counts the number of times the patient can sit down and stand up in 30 seconds. This test evaluates lower limb strength and it is associated to the cardiovascular capacity of elderly people.
Change from baseline in Berg Balance Scale at 16 weeks | from date to randomization at 16 weeks
  Berg Balance Scale (BERG) is composed by 14 tasks related to daily life and each item has one ordinal scale of five alternatives which vary from 0 to 4 points, with a total of 56 points.
Change from baseline in Trail Making Test at 16 weeks | from date to randomization at 16 weeks
  Both parts of the Trail Making Test consist of 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1 - 13) and letters (A - L); as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters. The patient should be instructed to connect the circles as quickly as possible, without lifting the pen or pencil from the paper.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil